CLINICAL TRIAL: NCT07266415
Title: A 2-Week, Single-Center, Double-blind, Exploratory Study to Evaluate the Safety and Efficacy of the Sleep Inducing Digital Sound Application on Pregnant Women in Their 1st and 2nd Trimester With Insomnia
Brief Title: Study for Pregnant Women With Insomnia Using Sleep Inducing Digital Sound Application
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: BELL Therapeutics Inc. (Industry)
Responsible Party: Principal Investigator, Jee Yoon Park, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-2501-950-302
Record Dates: First submitted 2025-04-20; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-06

CONDITIONS: Insomnia; Pregnancy, First Trimester; Pregnancy, Second Trimester
Keywords: insomnia; pregnancy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental)
  Interventions: Device: Sleep inducing digital sound application
- Sham-controlled group (Sham Comparator)
  Interventions: Device: Provides meaningless sound in application
- Control group (Placebo Comparator): Sleep Hygiene Education in application
  Interventions: Device: Provides Sleep hygiene education text in application

INTERVENTIONS:
Device: Sleep inducing digital sound application — Application: BELL-001
  Arms: Experimental group
Device: Provides meaningless sound in application — Sham application intervention
  Arms: Sham-controlled group
Device: Provides Sleep hygiene education text in application — Placebo application
  Arms: Control group

SUMMARY:
This study aims to evaluate the safety and efficacy of sleep inducing digital sound application on pregnant women in their 1st and 2nd trimester with insomnia

DETAILED DESCRIPTION:
Duration of study period (per participant): Screening period (0-1 week), Intervention period (2 weeks), Follow-up period (1 week, without digital application use). Patient needs to visit the site at least 1 time (Screening). Other procedures will be conducted online. First visit is before the screening period, mainly to on-board patients and to train patients for accurate usage of the digital application.

ELIGIBILITY:
Inclusion Criteria:

* 19 years older
* pregnant women in their 1st and 2nd trimester
* suffering from insomnia symptom
* scored 10 or high in screening ISI
* a person who voluntarily agreed to participate in this RCT

Exclusion Criteria:

* Has a confirmed diagnosis of insomnia disorder other than chronic insomnia based on DSM-5(ex. Narcolepsy, Periodic Limb Movement, Restless Leg syndrome, etc)
* Has a confirmed diagnosis of other neuropsychiatric disease
* Has an history of suicidal ideat or attempt
* Shift worker
* Going through other interventions regarding insomnia(sleeping pills, light therapy, other alternative interventions)
* Has a severe auditory, visual, or cognitive impairment
* A person who cannot familiarize with the usage of smartphones and digital applications
* Has a history of alcohol or other substance use disorder
* A person with high risk pregnancy considered inadequate to participate in this trial by obstetric experts
* A person considered inadequate to participate in this trial by a clinical expert

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-03-18 (Estimated); Study Completion 2026-05-18 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measurement | 1 week
  Insomnia severity index

SECONDARY OUTCOMES:
Sleep Latency (SL, Minutes), assessed using a sleep diary | 1 week
Sleep Latency (SL, Minutes), assessed using a smartwatch | 1 week
Sleep Efficiency (SE, Percentage), assessed using a sleep diary | 1 week
Sleep Efficiency (SE, Percentage), assessed using a smartwatch | 1 week
Wake After Sleep Onset (WASO, Minutes), assessed using a sleep diary | 1 week
Wake After Sleep Onset (WASO, Minutes), assessed using a smartwatch | 1 week
Total Sleep Time (TST, Minutes), assessed using a sleep diary | 1 week
Total Sleep Time (TST, Minutes), assessed using a smartwatch | 1 week
Sleep Quality (SQ, Score 1-10; bad-good), assessed using a sleep diary | 1 week
Pittsburgh Sleep Quality Index (PSQI, Score 0-21; better-worse) | 2 weeks
Edinburgh Postnatal Depression Scale (EPDS, Score 0-30; better-worse) | 2 weeks
Generalized Anxiety Disorder-7 (GAD-7, Score 0-21; better-worse) | 2 weeks
Pregnancy-Related Anxiety Questionnaire (PRAQ, Score 32-128; better-worse) | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea